CLINICAL TRIAL: NCT00123916
Title: Benznidazole Evaluation for Interrupting Trypanosomiasis - The BENEFIT Trial
Brief Title: BENEFIT: Evaluation of the Use of Antiparasital Drug (Benznidazole) in the Treatment of Chronic Chagas' Disease
Acronym: BENEFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); World Health Organization (Other); Instituto Dante Pazzanese de Cardiologia (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Salim Yusuf's office, Principal Co-Investigator, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEN01; CONEP-11394 (Other: Comissão Nacional de Ética em Pesquisa (CONEP))
Record Dates: First submitted 2005-07-21; First posted 2005-07-26 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Chagas Disease; Trypanosomiasis; Heart Disease
Keywords: Chagas Disease; Trypanosomiasis; Benznidazole; Chronic Heart disease; Trypanosoma Cruzi
MeSH Terms: conditions — Chagas Disease; Trypanosomiasis; Heart Diseases | interventions — benzonidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benznidazole (Experimental): 40 - 80 days (according to body weight) treatment with benznidazol
  Interventions: Drug: Benznidazole
- Placebo (Placebo Comparator): 40 - 80 days (according to body weight) treatment with matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benznidazole — Daily po Benznidazole or placebo (weight based) during 40 - 80 days (depending on body weight)
  Other Names: Rochagan/LaFepe
  Arms: Benznidazole
Drug: Placebo — a dose calculated as 5mg/kg/day for 60 days, now administered as a fixed daily dose of 300mg during 40 - 80 days of treatment - period adjusted according to the patient's body weight to a total minimum dose of 12g (corresponding to 40kg) and a total maximum dose of 24g (corresponding to 80kg)
  Other Names: Rochagan/LaFepe
  Arms: Placebo

SUMMARY:
Evaluate if benznidazole, an antiparasite drug, given at a dose calculated as 5mg/kg/day for 60 days, now administered as a fixed daily dose of 300mg during 40 to 80 days of treatment - period adjusted according to the patient's body weight to a total minimum dose of 12g (corresponding to 40kg) and a total maximum dose of 24g (corresponding to 80kg) - reduces morbidity and mortality in patients with Chronic Chagas' Cardiomyopathy (CCC).

The BENEFIT study is being conducted by the Population Health Research Institute (in Hamilton, Canada) and the Institute Dante Pazzanese de Cardiologia (Sao Paulo, Brazil) together with a Steering Committee, and an independent Safety Monitoring Board.

DETAILED DESCRIPTION:
A randomized double-blind controlled clinical trial investigating the role of benznidazole in patients with chronic Chagas' heart disease.

Chagas disease has 3 phases: acute, undetermined and chronic phases. There are no clinical trials up to date that have investigated the use of antiparasitic drugs in patients that are in the chronic phase.

This study will evaluate the efficacy and safety of benznidazole (an antiparasitic drug) in patients with chronic Chagas' heart disease. Evaluate if benznidazole, an antiparasite drug, given at a dose calculated as 5mg/kg/day for 60 days, now administered as a fixed daily dose of 300mg during 40 to 80 days of treatment - period adjusted according to the patient's body weight to a total minimum dose of 12g (corresponding to 40kg) and a total maximum dose of 24g (corresponding to 80kg) - reduces morbidity and mortality in patients with Chronic Chagas' Cardiomyopathy (CCC). It will be developed in 49 study centres in Argentina, Bolivia,Brazil,Colombia, and El Salvador - countries with high incidence of Chagas Disease.

The Pilot study is evaluating if benznidazole is effective in producing parasitic cure (PCR negativization or reducing parasitic load) in chronic Chagas Disease as well as assessing the feasibility of conducting a large trial in chronic Chagas Disease in South America.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients (between 18 and 75 years of age) with serological evidence of Chagas infection (any combination of 2 positive tests) and that have one or more of the following:
* Abnormal electrocardiogram with at least two components (complete RBBB or LBBB; left anterior or posterior fascicular block; ventricular premature beat; first degree atrioventricular [AV] block; Mobitz type I AV block; sinus bradycardia; primary ST-T changes; abnormal Q waves; low voltage QRS; or atrial fibrillation);
* Abnormal ECG (Mobitz type II, advanced or third degree AV block);
* Increased cardiothoracic ratio (> 0.50);
* Complex ventricular arrythmias on 24 hour ambulatory ECG monitoring;
* Evidence of regional wall motion abnormality or reduced global left ventricular systolic function or increased left ventricular and diastolic diameter on 2D-Echo.

Exclusion Criteria:

Patients will be excluded if having:

* NYHA heart failure class IV or decompensated heart failure
* Evidence of concomitant coronary artery disease (CAD) or other etiology of dilated cardiomyopathy
* Previous treatment with antitrypanosomal agents or an accepted indication for antiparasitic therapy
* Inability to comply with follow-up visits
* History of severe alcohol abuse within 2 years
* Known chronic renal or hepatic insufficiency or hepatic insufficiency
* Pregnancy or breast feeding
* Megaesophagus with swallowing impairment
* Other severe disease significantly curtailing life expectancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2854 (Actual)
Dates: Start 2004-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Composite of First of cardiovascular events: Death, Resuscitated Cardiac Arrest, Sustained VentricularTachycardia, New/worsening Heart Failure, New Pacemaker/ICD, Stroke/TIA or other Embolic Events, Cardiac Transplant. | through study completion, an average of 5 years
  Composite cardiovascular outcome,

SECONDARY OUTCOMES:
New development of any of the following echo changes, segmental wall motion abnormalities, ventricular aneurysm, reduction in LV ejection fraction >5%, increase in LVDD> 5 mm compared to baseline. | through study completion, an average of 5 years
New 12 lead ECG alterations (complete bundle branch block, fascicular block, advanced atrio-ventricular block, atrial fibrillation, etc). | through study completion, an average of 5 years
Progression of NYHA functional class by at least one category | through study completion, an average of 5 years
New 12 lead electrocardiogram (ECG) alterations (complete bundle branch block; fascicular block, advanced atrio-ventricular block, atrial fibrillation, etc.) | through study completion, an average of 5 years
Progression of New York Heart Association (NYHA) functional class by at least one category | through study completion, an average of 5 years
Evaluation of safety (adverse events: dermatitis, peripheral neuropathy, gastro-intestinal intolerance, leucopenia [2500 x 10^9 L]), tolerance and adherence to treatment | through study completion, an average of 5 years
Determination of the efficacy of benznidazole in patients with Chronic Chagas heart disease based on a 50% reduction in both qualitative and quantitative PCR. | through study completion, an average of 5 years
  Polymerase Chain Reaction study on patient's blood samples and report negativization at the end of treatment, 2Y and final visit.
Safety and tolerability of benznidazole | through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Morillo, MD, Study Chair — Population Health Research Institute - McMaster University; Jose Antonio Marin-Neto, MD, PhD, Study Chair — University of Sao Paulo; Salim Yusuf, MD, DPh, Study Chair — Population Health Research Institute - McMaster University; Sergio Sosa-Estani, MD, PhD, Principal Investigator — Argentina National Coordinator - CenDIE, Argentina; Fernando Rosas, M.D., Principal Investigator — Fundacion Clinica Shaio, Bogota, Colombia
Locations (36):
- Argentina (17):
  - BENEFIT Ivestigational Site, Buenos Aires, Apital Federal
  - BENEFIT Investigational Site, Belén de Escobar, Buenos Aires
  - BENEFIT Investigational Site, Isidro Casanova, Buenos Aires
  - BENEFIT Investigational Site, San Juan, Buenos Aires
  - BENEFIT Investigational Site, Santiago Del Estero, Buenos Aires
  - BENEFIT Investigational Site, Buenos Aires, Buenos Aires F.D.
  - BENEFIT Investigational Site, Catamarca, Catamarca Province
  - BENEFIT Investigational Site, Charata, Chaco Province
  - BENEFIT Investigational Site, Paraná, Entre Ríos Province
  - BENEFIT Investigational Site, Buenos Aires, General Rodríguez Partido
  - BENEFIT Investigational Site, San Salvador de Jujuy, Jujuy Province
  - BENEFIT Investigational Site, Corrientes, Rosario, Santa Fe
  - BENEFIT Investigational Site, Rosario, Santa Fe Province
  - BENEFIT Investigational Site, Añatuya, Santiago del Estero Province
  - BENEFIT Investigational Site, Santiago del Estero, Sgo. Del Estero
  - BENEFIT Investigational Site, Buenos Aires
  - BENEFIT Investigational Site, Salta
- BENEFIT Investigational Site, Tupiza, Potosí Department, Bolivia
- Brazil (15):
  - BENEFIT Investigational Site, Salvador, Bahaia
  - BENEFIT Investigational Site, Carmo, Belo Horizonte
  - BENEFIT Investigational Site, Brasília, Brazilian Federal District
  - BENEFIT Investigational Site, Goiânia, Goiás
  - BENEFIT Investigational Site, Uberaba, Minas Gerais
  - BENEFIT Investigational Site, Uberlândia, Minas Gerais
  - BENEFIT Investigational Site, Curitiba, Paraná
  - BENEFIT Investigational Site, Recife, Pernambuco
  - BENEFIT Investigational Site, Pelotas, Rio Grande do Sul
  - BENEFIT Investigational Site, Campinas, São Paulo
  - BENEFIT Investigational Site, Ribeirão Preto, São Paulo
  - BENEFIT Investigational Site, São José do Rio Preto, São Paulo
  - BENEFIT Investigational Site, Votuporanga, São Paulo
  - BENEFIT Investigational Site, Rio de Janeiro
  - BENEFIT Investigational Site, São Paulo
- Colombia (2):
  - BENEFIT Investigational Site, Bogotá, Bogota D.C.
  - BENEFIT Investigational Site, San Gil, Santander Department
- BENEFIT Ivestigational Site, San Salvador, El Salvador

REFERENCES:
- [Background] Marin-Neto JA, Rassi A Jr, Morillo CA, Avezum A, Connolly SJ, Sosa-Estani S, Rosas F, Yusuf S; BENEFIT Investigators. Rationale and design of a randomized placebo-controlled trial assessing the effects of etiologic treatment in Chagas' cardiomyopathy: the BENznidazole Evaluation For Interrupting Trypanosomiasis (BENEFIT). Am Heart J. 2008 Jul;156(1):37-43. doi: 10.1016/j.ahj.2008.04.001. PMID 18585495
- [Derived] Morillo CA, Marin-Neto JA, Avezum A, Sosa-Estani S, Rassi A Jr, Rosas F, Villena E, Quiroz R, Bonilla R, Britto C, Guhl F, Velazquez E, Bonilla L, Meeks B, Rao-Melacini P, Pogue J, Mattos A, Lazdins J, Rassi A, Connolly SJ, Yusuf S; BENEFIT Investigators. Randomized Trial of Benznidazole for Chronic Chagas' Cardiomyopathy. N Engl J Med. 2015 Oct;373(14):1295-306. doi: 10.1056/NEJMoa1507574. Epub 2015 Sep 1. PMID 26323937
- [Derived] Marin-Neto JA, Rassi A Jr, Avezum A Jr, Mattos AC, Rassi A, Morillo CA, Sosa-Estani S, Yusuf S; BENEFIT Investigators. The BENEFIT trial: testing the hypothesis that trypanocidal therapy is beneficial for patients with chronic Chagas heart disease. Mem Inst Oswaldo Cruz. 2009 Jul;104 Suppl 1:319-24. doi: 10.1590/s0074-02762009000900042. PMID 19753491
- See also: Population Health Research Institute — http://www.phri.ca
- See also: Instituto Dante Pazzanese de Cardiologia — http://www.idpc.org.br/pesquisa/